CLINICAL TRIAL: NCT03664778
Title: Cancer Detection Rate of Abbreviated (Fast) Breast MRI (AB-MR) After Negative Digital Breast Tomosynthesis in Women Status Post Conservation Therapy (BCT)
Brief Title: Abbreviated Breast MRI After Cancer Treatment
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 829400
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
500 patients will be prospectively recruited to undergo a fast breast MRI examination. The women will be recruited for the study will meet the following criteria: 1. status post primary breast cancer treated with breast conservation therapy 3 years prior to recruitment 2. negative DBT examination six months prior to recruitment 3. all breast densities 4. clinically asymptomatic - no palpable masses, focalthickening, or clinically significant discharge We will identify these patients EPIC database utilizing the date of their last mammogram. The patients will be sent a letter explaining the study and the opportunity to enroll in the study. Interested patients may contact our research coordinators by the phone number provided in the letter. The study recruitment information will also be shared with referring physicians. Physicians may also directly refer patients to the study.

DETAILED DESCRIPTION:
Women treated for primary breast cancer who undergo breast conservation therapy face an increased risk of developing a second breast cancer in the ipsilateral and the contralateral breast. Although mammographic screening is recommended annually, the sensitivity of mammography is limited in these patients due to the post treatment changes from previous surgery and radiation. We propose supplemental screening with an abbreviated form of breast MRI ("fast MRI") examination in addition to mammographic screening, in order to study whether we can detect subclinical disease that may not be detected on mammography or on physical examination. Several tumor characteristics correlate with overall survival such as the extent of local recurrence and the size of the local recurrence, with larger extent and increased size of local recurrence correlating with adverse survival. In addition, the shorter time interval to the ipsilateral breast cancer recurrence from completion of treatment, is associated with increased risk of developing distant metastasis and breast cancer mortality. We will assess additional cancer detection with fast MRI after negative mammography in the ipsilateral as well as the contralateral breast. The goal of the supplemental screening with fast breast MRI would be to detectsubclinical disease not detected on mammography and thus improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Status post primary breast cancer (both invasive and DCIS) treated with breast conservation therapy at least three years prior to recruitment
2. Negative DBT examination within six months prior to recruitment
3. All breast densities
4. Clinically asymptomatic - no palpable masses or focal thickening, etc.

Exclusion Criteria:

1. Patients who are pregnant or lactating.
2. Patients who have not had a mammogram (digital breast tomosynthesis) in the past 6 months.
3. Patients who are unwilling or unable to provide written informed consent.
4. Patients symptomatic for breast disease (e.g. experiencing discharge, lumps, etc.).
5. Recent breast surgery in the past two years including breast enhancements (e.g. implants or injections) benign surgical biopsies.
6. Patients who are unable to receive an MRI with Gadolinium contrast.
7. Patients who have not had an MRI of the breast within the past year.

Ages: 18 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who have had primary breast cancer treated with breast conservation therapy and who fit the inclusion criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Invasive breast cancer detection | 4 years
  To detect subclinical disease not detected on mammography

SECONDARY OUTCOMES:
DCIS and invasive cancer detection rate | 4 years
  To detect DCIS/Cancer not detected on mammography
Tumor size | 4 years
  Tumor size
Axillary nodal status | 4 years
  Axillary nodal status
Time to recurrence | 4 years
  To determine the time of recurrence
Ipsilateral and contralateral breast cancer detection | 4 years
  Ipsilateral and contralateral breast cancer detection

CONTACTS AND LOCATIONS:
Overall Officials: Susan Weinstein, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- UPenn, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No